CLINICAL TRIAL: NCT01261845
Title: Ecology of Medical Care - Utilisation of Health Care in Austria
Acronym: ECOHCARE
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Otto Pichlhoefer, MD, Medical University of Vienna
Other Study IDs: 13683; 13575 (Other: Oesterreichische Nationalbank)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Health Behavior
Keywords: Delivery of Health Care; Equity in Health Services; Ethnic Groups; Health Services Research; Health Surveys; Immigration; Referral and Consultation; Resource Allocation; Social Justice; Vulnerable Populations
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
BACKGROUND: A proper understanding of the attitudes towards its own health status and concise estimates concerning the health seeking behavior of the different subgroups of a population are highly desirable. The structure of the Austrian population with regard to its age distribution and the proportion of people with immigrant backgrounds have been rapidly changing in recent years. Questions of allocating limited resources and meeting the needs of under-served populations have become increasingly important. However, data that could illuminate these issues are sparse and therefore obtaining them will be important for making sensible policy decisions.

METHODS: A telephone survey of the Austrian population for the assessment of the occurrence of any health complaint and the subsequent help seeking behavior with special emphasize on under-served minority groups - migrant population, elder people, and female gender.

AIMS: Our analysis of the data obtained should help to clarify some hitherto undocumented aspects and should provide the evidence for building a better health care infrastructure with equality of access and efficient coordination. We also hope that this information can help to allocate resources strategically according to needs and cost-efficiency in health care.

ELIGIBILITY:
Inclusion Criteria:

* 15 years and older

Exclusion Criteria:

* younger than 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Austrian population 15 years and older .
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of health complaints | 1 month
  The occurrence of any health complaint and the subsequent help seeking behaviour with special emphasis on under-served minority groups.
Prevalence of dysphoric disorders | 2 weeks
  The prevalence of depression and GAD will be assessed by the PHQ-2 and GAD-2 respectively.

SECONDARY OUTCOMES:
Utilization of CAM | 1 month
  The utilization of CAM and a classification scheme for CAM methods in Austria.
Utilization of Health Care Resources in Austria | 1 month
  The utilization of health care resources of the Austrian population with respect to Primary, Secondary and Tertiary levels of care.
Case vignettes for calibration of response measures | 1 month
  The use of case vignettes to calibrate response measures across various ethnic minority groups.

CONTACTS AND LOCATIONS:
Overall Officials: Otto Pichlhoefer, MD, Principal Investigator — MedUni Vienna
Locations (1):
- Department for General Practice and Family Medicine, Center for Public Health at the Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Pichlhofer O, Maier M. Unregulated access to health-care services is associated with overutilization--lessons from Austria. Eur J Public Health. 2015 Jun;25(3):401-3. doi: 10.1093/eurpub/cku189. Epub 2014 Nov 23. PMID 25417940